CLINICAL TRIAL: NCT01688687
Title: The Accuracy of Probe-based Confocal Endomicroscopy Versus Conventional Biopsies for the Diagnosis of Superficial Gastric Neoplasias
Brief Title: Conventional Biopsies vs pCLE for Diagnosis of Superficial Gastric Neoplasia
Acronym: pCLE
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Gene Hyun Bok, M.D., Soonchunhyang University Hospital
Other Study IDs: MD-2012-01
Record Dates: First submitted 2012-09-06; First posted 2012-09-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Early Gastric Cancer; Gastric Dysplasia
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endscopic resection specimens of gastric neoplasia. Speciments were obtained either by endoscopic mucosal resection or endoscopic submucosal dissection.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Superficial gastric neoplasia: Patients with superficial gastric neoplasia on diagnostic endoscopy, recieved both conventional endoscopic forcpes biopsies and pCLE. All patients were subject to endoscopic resection of the lesion.
  Interventions: Procedure: Endoscopic submucosal dissection

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection

SUMMARY:
Confocal endomicroscopy (CLE) allows real-time in-vivo high-resolution and high-magnification imaging of the gastrointestinal epithelium, which is comparable to histopathology. Previous studies have investigated the accuracy of pCLE for diagnosis and differentiated of colorectal polyps, Barrett's esophagus and pancreaticobiliary strictures. However, to date there are limited data exploring the application of pCLE to gastric lesions, and this is the first study comparing the diagnosis of conventional forceps biopsy with that of pCLE using the final specimens obtained from endoscopic resection as a reference standard. The aims of this study were (1) the accuracy of pCLE compared to conventional forceps biopsy using histopathology results following endoscopic resection as a reference, and (2) comparison of "real time" in-vivo pCLE diagnosis with that of blinded "off-line" pCLE diagnosis, and off-line interobserver agreement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biospy proven superficial gastric neoplasia, suitable for endoscopic resection.

Exclusion Criteria:

* Patients with uncorrectable coagulopathy,
* liver cirrhosis,
* acute gastrointestinal bleeding,
* pregnancy,
* breast feeding,
* documented allergy to fluorescein,
* patients with lesions that were deemed unsuitable for endoscopic resection, and
* patients without documented conventional biopsy results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to a tertiary medical center for endoscopic resection of gastric superficial lesions.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The accuracy of pCLE compared to conventional forceps biopsy | in-vivo pCLE accuracy compared to conventional forceps biopsy was assessed 1-2 weeks prior to endoscopic resection.
  The accuracy of pCLE compared to conventional forceps biopsy was assessed using histopathology results following endoscopic resection as a reference

SECONDARY OUTCOMES:
Comparison of "real time" in-vivo pCLE diagnosis with that of blinded "off-line" pCLE diagnosis. | 1-3 months after endoscopic resection and final histopathological analysis
Off-line pCLE interobserver agreement | 1-3 months after endoscopic resection and final histopathological analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Soonchunhyang University Seoul Hospital, Seoul, South Korea

REFERENCES:
- [Result] Wallace M, Lauwers GY, Chen Y, Dekker E, Fockens P, Sharma P, Meining A. Miami classification for probe-based confocal laser endomicroscopy. Endoscopy. 2011 Oct;43(10):882-91. doi: 10.1055/s-0030-1256632. Epub 2011 Aug 4. PMID 21818734
- [Result] Jeon SR, Cho WY, Jin SY, Cheon YK, Choi SR, Cho JY. Optical biopsies by confocal endomicroscopy prevent additive endoscopic biopsies before endoscopic submucosal dissection in gastric epithelial neoplasias: a prospective, comparative study. Gastrointest Endosc. 2011 Oct;74(4):772-80. doi: 10.1016/j.gie.2011.05.005. Epub 2011 Jul 29. PMID 21802680
- [Result] Shahid MW, Buchner AM, Raimondo M, Woodward TA, Krishna M, Wallace MB. Accuracy of real-time vs. blinded offline diagnosis of neoplastic colorectal polyps using probe-based confocal laser endomicroscopy: a pilot study. Endoscopy. 2012 Apr;44(4):343-8. doi: 10.1055/s-0031-1291589. Epub 2012 Mar 1. PMID 22382851
- [Result] Wallace MB, Crook JE, Saunders M, Lovat L, Coron E, Waxman I, Sharma P, Hwang JH, Banks M, DePreville M, Galmiche JP, Konda V, Diehl NN, Wolfsen HC. Multicenter, randomized, controlled trial of confocal laser endomicroscopy assessment of residual metaplasia after mucosal ablation or resection of GI neoplasia in Barrett's esophagus. Gastrointest Endosc. 2012 Sep;76(3):539-47.e1. doi: 10.1016/j.gie.2012.05.004. Epub 2012 Jun 28. PMID 22749368
- [Result] Kuiper T, Kiesslich R, Ponsioen C, Fockens P, Dekker E. The learning curve, accuracy, and interobserver agreement of endoscope-based confocal laser endomicroscopy for the differentiation of colorectal lesions. Gastrointest Endosc. 2012 Jun;75(6):1211-7. doi: 10.1016/j.gie.2012.01.040. Epub 2012 Mar 28. PMID 22459661